CLINICAL TRIAL: NCT02964494
Title: The Congenital Dyserythropoietic Anemia Registry (CDAR)
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-2727_CDAR
Record Dates: First submitted 2016-10-04; First posted 2016-11-16 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Congenital Dyserythropoietic Anemia (CDA)
MeSH Terms: conditions — Anemia, Dyserythropoietic, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Subject DNA isolated from subject's oral cells or blood or other biological samples donated to be used for gene sequencing diagnostic studies (evaluate for known or novel genes that may be causative of CDA)
  Bone marrow will be collected ONLY when bone marrow samples are being collected for standard diagnostic or treatment related reasons. No interventional procedure other than a voluntary blood draw, if patient consents, is required as part of the CDAR Registry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators have created and maintain a comprehensive registry for patients with the diagnosis of Congenital Dyserythropoietic Anemia (CDA) in North America. The goal of this registry is to collect long-term confidential data on patients with CDA in the US, Canada, and Mexico and maintain a bio-repository of de-identified patient blood and bone marrow specimens as a tool for the investigation of epidemiology, natural history, biology, and molecular pathogenetic mechanisms of CDA.

DETAILED DESCRIPTION:
We have established and maintain a CDA registry (CDAR): a comprehensive registry of subjects with the diagnosis of any type of congenital dyserythropoietic anemia in North America. Subjects and their physicians have expressed interest in participating in a national/international registry that could promote research and further understanding of this rare disease-group.

CDAs consist a heterogeneous group of rare genetic disorders causing ineffective erythropoiesis with the characteristic finding of multinuclear erythroid precursors in the bone marrow. The other hematopoietic lineages seem unaffected. The diagnosis of CDA is clinically challenging and is based on identifying the characteristic morphology of erythroblasts in the bone marrow of subjects presenting with chronic anemia, frequently with evidence of hemolysis but suboptimal reticulocytosis, and iron overload. Three types are well-defined by marrow morphology, although a recent classification recognizes seven different genetic types. Since certain gene defects were identified in the different types of CDAs, our understanding of the biology and pathogenesis of these diseases has been improving. However, many gaps still exist in our understanding of the related molecular mechanisms primarily due to the rarity of the disease and the lack of systematic approach to study these subjects. In addition, the heterogeneity observed among subjects and the clinical overlap with other hematologic disorders, namely hemolytic anemias with brisk erythropoietic response that may be associated with erythroid dysplasia, and with ineffective erythropoiesis, further complicates the diagnosis and often delays appropriate diagnosis and therapy.

The purpose of CDAR is to maintain a database and bio-repository for patients with CDA and their families in order to systematically study this rare disease-group. Data regarding these subjects are collected confidentially at initial presentation or diagnosis and periodically thereafter over a long period of time (>15 years). In addition, blood, bone marrow (only if that procedure is clinically indicated based on the primary hematologist's decision) and/or DNA samples of enrolled subjects are stored for research studies with the aim to improve our understanding, diagnosis, and treatment of CDA.

The study continues recruiting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Congenital Dyserythropoietic Anemia (CDA), whether a genetic mutation is identified or not
* Evidence of congenital anemia/jaundice or a positive family history
* Evidence of ineffective erythropoiesis
* Typical morphological appearance of bone marrow erythroblasts
* All ages (ages 0-99)

Exclusion Criteria:

* Diagnosis of cancer
* Myelodysplasia
* Secondary dyserythropoiesis: e.g.; vitamin B12 deficiency or drug-related.

Note1: Patients with rare band 3 (SLC4A1) mutations recently described to be associated with dyserythropoiesis will be eligible since the mechanisms appear to involve direct participation of band 3 in the erythroblast mitosis and cytokinesis.

Note2: Siblings, parents, and family members of patients with confirmed CDA diagnosis are encouraged to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Congenital Dyserythropoietic Anemia (CDA)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-08-29 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Age and symptoms at presentation and/or diagnosis | From study entry to >15 years
  Clinical and laboratory information will be collected by the patient and the referring physician with questionnaires in order to obtain the natural history of the disease, including correlations, epidemiology, and biology of the different types of CDA.
Degree of anemia | From study entry to >15 years
  Clinical and laboratory information will be collected by the patient and the referring physician with questionnaires in order to obtain the natural history of the disease, including correlations, epidemiology, and biology of the different types of CDA.
Clinical course during | From study entry to >15 years
  infancyClinical and laboratory information will be collected by the patient and the referring physician with questionnaires in order to obtain the natural history of the disease, including correlations, epidemiology, and biology of the different types of CDA.
Growth and development, endocrinologic evaluation, skeletal | From study entry to >15 years
  dysplasiasClinical and laboratory information will be collected by the patient and the referring physician with questionnaires in order to obtain the natural history of the disease, including correlations, epidemiology, and biology of the different types of CDA.
Transfusion requirements | From study entry to >15 years
  requirementsClinical and laboratory information will be collected by the patient and the referring physician with questionnaires in order to obtain the natural history of the disease, including correlations, epidemiology, and biology of the different types of CDA.
Evidence and complications of hemolysis and of extramedullary | From study entry to >15 years
  erythropoiesisClinical and laboratory information will be collected by the patient and the referring physician with questionnaires in order to obtain the natural history of the disease, including correlations, epidemiology, and biology of the different types of CDA.
Iron overload, frequency and methods of monitoring, iron chelators, effectiveness and history of side effects if | From study entry to >15 years
  usedClinical and laboratory information will be collected by the patient and the referring physician with questionnaires in order to obtain the natural history of the disease, including correlations, epidemiology, and biology of the different types of CDA.
Splenomegaly, history of splenectomy and effect if performed; possible complications, e.g. thrombosis or | From study entry to >15 years
  sepsisClinical and laboratory information will be collected by the patient and the referring physician with questionnaires in order to obtain the natural history of the disease, including correlations, epidemiology, and biology of the different types of CDA.
History of stem cell transplant, effect, complications | From study entry to >15 years
  Clinical and laboratory information will be collected by the patient and the referring physician with questionnaires in order to obtain the natural history of the disease, including correlations, epidemiology, and biology of the different types of CDA.
Other medications, e.g. interferon A for CDA-I, effect on anemia and on transfusion frequency, any side effects | From study entry to >15 years
  notedClinical and laboratory information will be collected by the patient and the referring physician with questionnaires in order to obtain the natural history of the disease, including correlations, epidemiology, and biology of the different types of CDA.
Ethnic background and demographic information will also be collected for epidemiologic studies | From study entry to >15 years
  Clinical and laboratory information will be collected by the patient and the referring physician with questionnaires in order to obtain the natural history of the disease, including correlations, epidemiology, and biology of the different types of CDA.

CONTACTS AND LOCATIONS:
Overall Officials: Theodosia Kalfa, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data regarding subjects that meet inclusion will be collected confidentially at initial presentation or diagnosis and periodically thereafter over a long period of time (>15 years). In addition, blood, bone marrow and/or DNA samples of enrolled subjects will be stored for research studies with the aim to improve diagnosis, treatment and care of CDA.
  The samples and medical information (that is not associated with a patient's name) may be used by other researchers studying CDA, at Cincinnati Children's Hospital Medical Center or at other institutions. The researchers must get Institutional Review Board (a board that is in charge of regulating research done on people) approval prior to requesting data and/or samples from this repository if applicable. No identifying information (that associates the medical information with the subject or sample) will be available to them.

REFERENCES:
- [Background] Seu KG, Trump LR, Emberesh S, Lorsbach RB, Johnson C, Meznarich J, Underhill HR, Chou ST, Sakthivel H, Nassar NN, Seu KJ, Blanc L, Zhang W, Lutzko CM, Kalfa TA. VPS4A Mutations in Humans Cause Syndromic Congenital Dyserythropoietic Anemia due to Cytokinesis and Trafficking Defects. Am J Hum Genet. 2020 Dec 3;107(6):1149-1156. doi: 10.1016/j.ajhg.2020.10.013. Epub 2020 Nov 12. PMID 33186543
- [Background] Boucher AA, Dayton VJ, Pratt AR, Nassar NN, Elgammal Y, Kalfa TA. Three-generation female cohort with macrocytic anemia and iron overload. Am J Hematol. 2025 Jan;100(1):133-138. doi: 10.1002/ajh.27489. Epub 2024 Sep 27. No abstract available. PMID 39329459
- [Background] Hernandez G, Romero-Cortadellas L, Ferrer-Cortes X, Venturi V, Dessy-Rodriguez M, Olivella M, Husami A, De Soto CP, Morales-Camacho RM, Villegas A, Gonzalez-Fernandez FA, Morado M, Kalfa TA, Quintana-Bustamante O, Perez-Montero S, Tornador C, Segovia JC, Sanchez M. Mutations in the RACGAP1 gene cause autosomal recessive congenital dyserythropoietic anemia type III. Haematologica. 2023 Feb 1;108(2):581-587. doi: 10.3324/haematol.2022.281277. No abstract available. PMID 36200420
- [Background] Yenwongfai LN, Arora R, Smith AP, Kalfa T, Husami A, Radulescu V, Myers K, Lorsbach R. Pediatric myelofibrosis due to compound heterozygous MPIG6B mutations in a patient of European ancestry. Pediatr Blood Cancer. 2023 Mar;70(3):e30023. doi: 10.1002/pbc.30023. Epub 2022 Oct 2. No abstract available. PMID 36184776
- [Background] Harms FL, Rexach JE, Efthymiou S, Aynekin B, Per H, Gulec A, Nampoothiri S, Sampaio H, Sachdev R, Stoeva R, Myers K, Pena LDM, Kalfa TA, Chard M, Klassen M, Pries M, Kutsche K. Loss of TBC1D2B causes a progressive neurological disorder with gingival overgrowth. Eur J Hum Genet. 2024 May;32(5):558-566. doi: 10.1038/s41431-024-01563-5. Epub 2024 Feb 19. PMID 38374468
- [Result] Niss O, Lorsbach RB, Berger M, Chonat S, McLemore M, Buchbinder D, McCavit T, Shaffer LG, Simpson J, Schwartz JH, Meznarich J, Emberesh M, Seu KG, Zhang W, Kalfa TA; CDAR consortium. Congenital dyserythropoietic anemia type I: First report from the Congenital Dyserythropoietic Anemia Registry of North America (CDAR). Blood Cells Mol Dis. 2021 Mar;87:102534. doi: 10.1016/j.bcmd.2020.102534. Epub 2020 Dec 24. PMID 33401150
- [Derived] Kim S, Khoriaty R, Li L, McClune M, Kalfa TA, Wu J, Peltier D, Fujiwara H, Sun Y, Oravecz-Wilson K, King RA, Ginsburg D, Reddy P. ER-to-Golgi transport and SEC23-dependent COPII vesicles regulate T cell alloimmunity. J Clin Invest. 2021 Jan 19;131(2):e136574. doi: 10.1172/JCI136574. PMID 33463537